CLINICAL TRIAL: NCT06102252
Title: Combination Chemotherapy of Paclitaxel and Carboplatin With or Without Anthracycline as Aneo Adjuvant Treatment in Advanced Endometrial Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Gamal Mahmoud, assistant lecteurer oncology department sohag univerisity hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-7-01MD
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Paclitaxel; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): will receive the TEC regimen: paclitaxel 150mg/m2 infused for 3 hours, epirubicin 50mg/m2 infused for 30 minutes, and carboplatin 4mg/ml/min for one hour on day 1 every 3 weeks.
  Interventions: Drug: Paclitaxel/epirubcin/carboplatin
- group B (Active Comparator): ) will receive a ddTC regimen: paclitaxel 80mg/m2 for 3 hours on day 1,8,15. Carboplatin AUC 5 over one hour on day 1 repeated at 3-week intervals
  Interventions: Drug: Paclitaxel/carboplatin
- group C (Active Comparator): : paclitaxel 175 mg/m2 over 3 hours infusion on day 1-carboplatin AUC 5 over 1 hour on day 1 at 3 weeks intervals
  Interventions: Drug: Paclitaxel/carboplatin

INTERVENTIONS:
Drug: Paclitaxel/epirubcin/carboplatin — adjuvant treatment in endometrial carcinoma
  Arms: group A
Drug: Paclitaxel/carboplatin — Dose dense paclitaxel/carboplatin
  Arms: group B; group C

SUMMARY:
Endometrial cancer, the most common gynecologic cancer worldwide, is steadily increasing in developed countries.The early-stage forms of endometrial cancer are usually highly curable by surgical treatment alone, whereas advanced stages require adjuvant interdictions such as radiotherapy and chemotherapy. Platinum and anthracycline drugs have long been used as standard adjuvant chemotherapy drugs for advanced and recurrent endometrial carcinomas. In one study, the standard combination adjuvant treatment with AP was found to be more effective as an adjuvant therapy than whole abdominal irradiation

ELIGIBILITY:
Inclusion Criteria:• Age group: Histologically diagnosed with primary endometrial carcinoma

* more than 20 years old.

  * Any histological type of endometrial carcinoma
  * Stage III, IV
  * Stage one I or II with one or more of the following factors:

    1. Histologic grade 3 endometroid carcinoma with myometrial invasion still within half of the myometrium
    2. histological grade 1,2 endometroid carcinomas with invasion of over half of myometrium
    3. cervical stromal invasion
    4. vascular invasion; or
    5. serous carcinoma, clear cell carcinoma, or undifferentiated carcinoma
  * performance status 0-2
  * adequate function of all major organs

Exclusion Criteria:

* • Pt has received prior radiation or chemotherapy.

  * Pt with sarcomatous component
  * Metastatic endometrial carcinoma
  * Other malignancy
  * Unfit patient for chemotherapy

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Completion rate of chemotherapy | 6 months
  6 cycles

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Colombo N, Creutzberg C, Amant F, Bosse T, Gonzalez-Martin A, Ledermann J, Marth C, Nout R, Querleu D, Mirza MR, Sessa C; ESMO-ESGO-ESTRO Endometrial Consensus Conference Working Group. ESMO-ESGO-ESTRO Consensus Conference on Endometrial Cancer: Diagnosis, Treatment and Follow-up. Int J Gynecol Cancer. 2016 Jan;26(1):2-30. doi: 10.1097/IGC.0000000000000609. PMID 26645990
- [Background] Bestvina CM, Fleming GF. Chemotherapy for Endometrial Cancer in Adjuvant and Advanced Disease Settings. Oncologist. 2016 Oct;21(10):1250-1259. doi: 10.1634/theoncologist.2016-0062. Epub 2016 Jul 13. PMID 27412393
- [Background] Fujiwara K, Egawa-Takata T, Ueda Y, Kimura T, Yoshino K, Fujita M, Miyatake T, Ohta Y, Kamiura S, Enomoto T, Kimura T. Investigating the relative efficacies of combination chemotherapy of paclitaxel/carboplatin, with or without anthracycline, for endometrial carcinoma. Arch Gynecol Obstet. 2012 May;285(5):1447-53. doi: 10.1007/s00404-011-2154-9. Epub 2011 Nov 30. PMID 22127553
- [Background] Randall ME, Filiaci VL, Muss H, Spirtos NM, Mannel RS, Fowler J, Thigpen JT, Benda JA; Gynecologic Oncology Group Study. Randomized phase III trial of whole-abdominal irradiation versus doxorubicin and cisplatin chemotherapy in advanced endometrial carcinoma: a Gynecologic Oncology Group Study. J Clin Oncol. 2006 Jan 1;24(1):36-44. doi: 10.1200/JCO.2004.00.7617. Epub 2005 Dec 5. PMID 16330675